CLINICAL TRIAL: NCT06936514
Title: Bilateral Cervical Deep Lymphatic Trunk Decompression Combined With Mid-Cervical Deep Lymph Node-External Jugular Vein Anastomosis for the Treatment of Alzheimer's Disease: A Randomized Controlled Clinical Trial
Brief Title: Clinical Study on Deep Cervical Lymphatic Trunk Decompression Combined With Mid-Cervical Deep Lymph Node-External Jugular Vein Anastomosis for Alzheimer's Disease Treatment
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Oriental Neurosurgery Evidence-Based-Study Team (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB2025-YX-099-01
Record Dates: First submitted 2025-03-22; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer's Disease
MeSH Terms: interventions — Amyloid beta-Protein Precursor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Surgical group) (Experimental): bilateral cervical deep lymphatic trunk decompression combined with mid-cervical deep lymph node-external jugular vein anastomosis
  Interventions: Procedure: Bilateral Cervical Deep Lymphatic Trunk Decompression Combined with Mid-Cervical Deep Lymph Node-External Jugular Vein Anastomosis for Alzheimer's Disease
- control group (No Intervention): Patients are not subject to surgical intervention, only medication is administered

INTERVENTIONS:
Procedure: Bilateral Cervical Deep Lymphatic Trunk Decompression Combined with Mid-Cervical Deep Lymph Node-External Jugular Vein Anastomosis for Alzheimer's Disease — This intervention involves a surgical approach that combines bilateral cervical deep lymphatic trunk decompression with mid-cervical deep lymph node-external jugular vein anastomosis (LVA) to enhance lymphatic drainage in Alzheimer's Disease (AD) patients. The aim is to reduce the accumulation of neurotoxic substances in the brain, potentially improving cognitive function by facilitating waste clearance via the lymphatic system. The procedure is intended to restore normal lymphatic flow, potentially slowing disease progression in AD patients who have moderate to severe cognitive impairment.
  Arms: Experimental group (Surgical group)

SUMMARY:
The aim of this study is to evaluate the feasibility, safety, and efficacy of bilateral deep cervical lymphatic trunk decompression combined with mid and deep cervical lymph node-extracervical vein anastomosis in the treatment of patients with Alzheimer's disease. The study seeks to explore new treatment options that may improve the quality of life for patients with Alzheimer's disease.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is a progressive neurodegenerative disorder characterized by memory loss, cognitive impairment, and behavioral changes, ultimately leading to the inability of patients to perform daily activities independently. Despite the availability of various pharmacological treatments aimed at alleviating the progression of the disease, current therapeutic approaches are unable to effectively delay or reverse the course of AD. Therefore, the treatment of Alzheimer's disease remains a significant challenge in the global medical community. This issue is particularly pressing in patients with moderate to severe AD, as existing therapies have limited efficacy, creating a critical need for novel treatment strategies.

The discovery of the brain's lymphatic system has opened new avenues for the treatment of neurodegenerative diseases, including Alzheimer's disease. Recent studies have shown that the meningeal lymphatic vessels play a crucial role in clearing waste products from the brain, including neurotoxins such as amyloid-beta, which accumulate in patients with AD. Dysfunction of this lymphatic drainage system has been implicated in the pathogenesis of Alzheimer's disease. This insight has spurred interest in enhancing lymphatic drainage as a potential therapeutic approach for AD.

Lymphatic-venous anastomosis (LVA) is a surgical technique traditionally used to treat lymphedema and other lymphatic drainage disorders. It involves surgically connecting lymphatic vessels to nearby veins, allowing lymph fluid to flow directly into the venous system. Studies have suggested that LVA may help improve lymphatic drainage in the brain and potentially reduce the accumulation of harmful substances associated with Alzheimer's disease, thereby slowing disease progression. This research aims to provide valuable insights into the potential of enhancing brain lymphatic drainage as a therapeutic strategy for Alzheimer's disease, potentially leading to significant breakthroughs in its treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50-80 years;
2. Meet the diagnostic criteria for AD in the Revised Criteria for the Diagnosis and Staging of Alzheimer's Disease (2024) published by the National Institute Aging and Alzheimer's Association (NIA-AA);
3. Presence of moderate-to-severe cognitive impairment with a Clinical Dementia Rating (CDR) score ≥2;
4. Stable use of medication for ≥1 month and no planned change in medication within 3 months of randomisation;
5. The patients and their families had been informed of the purpose, significance, expected effects and potential risks of the study and voluntarily participated in the study by providing biological samples and signing an informed consent form.

Exclusion Criteria:

1. Dementia caused by other reasons: vascular dementia, central nervous system infections (e.g. HIV, syphilis, etc.), Creutzfeldt-Jakob disease, Huntington's chorea and Parkinson's disease, dementia with Lewy bodies, dementia due to traumatic brain injury, other physical and chemical factors (e.g. drug intoxication, alcohol intoxication, carbon monoxide intoxication, etc.), important physical diseases (e.g. hepatic encephalopathy, pulmonary encephalopathy, etc.), intracranial occupying lesions (e.g. subdural haematoma, brain tumour), endocrine system lesions (e.g. thyroid disease, parathyroid disease), and vitamin deficiency or any other cause of dementia;
2. Presence of current serious or unstable medical conditions, including cardiovascular, hepatic, renal, gastrointestinal, respiratory, endocrine, neurological (except for cognitive impairment of AD origin), psychiatric, immunological or haematological disorders, and any other condition which, in the opinion of the investigator, may affect the results of the analyses in this study; or a life expectancy of <24 months;
3. Presence of a history of cancer within 5 years, with the exception of non-metastatic basal cell and/or squamous cell carcinoma of the skin, cervical carcinoma in situ, non-progressive prostate cancer, or other cancers with a low risk of recurrence or spread;
4. Subjects with a current diagnosis of any primary psychiatric disorder other than cognitive impairment of AD origin, which requires exclusion if, in the opinion of the Investigator, the presence of the psychiatric disorder or symptom may interfere with interpretation of the effects of the LVA, interfere with cognitive assessment, or interfere with the subject's ability to complete the study. Exclusion is required for subjects with a history of schizophrenia or other chronic psychiatric illness;
5. Subjects who, in the judgement of the investigator, are actively suicidal and therefore considered to be at significant risk of suicide;
6. Illiteracy or insufficient education to complete the scale assessment;
7. A history of alcohol or drug abuse (other than a history of smoking) in the 2 years prior to the screening visit;
8. A clinically significant history of multiple or severe drug allergies, significant atopic sensitivities, or severe post-treatment hypersensitivity reactions (including, but not limited to, erythema multiforme, linear IgA dermatosis, toxic epidermal necrolysis-relaxation, and/or exfoliative dermatitis);
9. Clinically significant abnormalities of clinical significance (as determined by the investigator) on physical or neurological examination, vital signs, ECG, or clinical laboratory findings at screening that may be detrimental to the subject, interfere with the study, or suggest evidence of other causes of dementia;
10. MRI results at screening that show evidence of significant abnormalities suggesting the presence of another potential etiology of progressive cognitive impairment or the presence of clinically significant findings which may compromise the subject's ability to safely participate in the study. For example, >2 infarct foci >2 cm in diameter; infarct foci in key areas such as thalamus, hippocampus, internal olfactory cortex, parafactory cortex, angular gyrus, cortex and other subcortical grey matter nuclei; and a Fazekas Scale grade of >2 on the Cerebral White Matter Impairment Scale (CWMIS);
11. Presence of any contraindication to MRI, including claustrophobia, or presence of prohibited metallic (ferromagnetic) implants/pacemakers;
12. Presence of contraindications to LVA surgery, such as the presence of severe infection at the surgical site, severe cardiac, pulmonary, hepatic, renal, or other systemic functional abnormalities that cannot tolerate general anaesthesia surgery;
13. Currently participating in a clinical trial involving other interventional clinical trials, or participating in any other type of medical research that is considered scientifically or medically incompatible with this study;
14. Other reasons that prevent completion of this study: e.g., lack of a stable caregiver;
15. Female subjects who are pregnant or planning to become pregnant;
16. is a member of the Research Centre staff and/or his/her immediate family directly related to this study. Immediate family is defined as a spouse, parent, child, or sibling, whether biologically or legally adopted.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in Alzheimer's disease Assessment Scale-Cognitive Subscale 14 (ADAS-Cog14) | From enrollment to the end of treatment at 3 days, 7 days, 1 month, 3 months.
  The Alzheimer's disease Assessment Scale-Cognitive Subscale 14 (ADAS-Cog 14) will be used to evaluate the general cognitive function. ADAS-Cog 14 ranges from 0 to 90, and higher value represents a worse outcome.
Change in amyloid deposit in brain | Baseline and 3 months after surgery
  Change from baseline as measured by amyloid positron emission tomography (PET) scan using centiloids. The centiloid scale anchor points are 0 and 100, where 0 represents a high-certainty amyloid negative scan and 100 represents the amount of global amyloid deposition found in a typical AD scan. A negative change indicates an improvement from baseline.

SECONDARY OUTCOMES:
Change in Clinical Dementia Rating Scale sum of the boxes (CDR-SB) | From enrollment to the end of treatment at 3 days, 7 days, 1 month, 3 months.
  The Clinical Dementia Rating Scale sum of the boxes (CDR-SB) will be used to evaluate the general cognitive function. CDR-SB ranges from 0 to 18, and higher value represents a worse outcome.
Change in Mini-mental State Examination (MMSE) | From enrollment to the end of treatment at 3 days, 7 days, 1 month, 3 months.
  The Mini-mental State Examination (MMSE) will be used to evaluate the general cognitive function. MMSE ranges from 0 to 30, and higher value represents a better outcome.
Change in Montreal Cognitive Assessment (MoCA) | From enrollment to the end of treatment at 3 days, 7 days, 1 month, 3 months.
  The Montreal Cognitive Assessment (MoCA) will be used to evaluate the general cognitive function. MoCA ranges from 0 to 30, and higher value represents a better outcome.
Change in Hamilton Depression Scale (HAMD) | From enrollment to the end of treatment at 3 days, 7 days, 1 month, 3 months.
  The Hamilton Depression Scale (HAMD) will be used to evaluate the general depression status. HAMD ranges from 0 to 52, and higher value represents a better outcome.
Chang in Hamilton Anxiety Scale (HAMA) | From enrollment to the end of treatment at 3 days, 7 days, 1 month, 3 months.
  The Hamilton Anxiety Scale (HAMA) will be used to assess general anxiety status.The HAMA ranges from 0 to 56, with higher values resulting in better outcomes.
Changes in AD-related biomarkers | From enrollment to the end of treatment at 3 days, 7 days, 1 month, 3 months.
  Change from baseline in blood levels of Aβ42, Aβ40, Aβ42/40, pTau217, and pTau181.

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Tianjin Medical University, 154 Anshan Road, Heping District, Tianjin, China, Tianjin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benveniste H, Liu X, Koundal S, Sanggaard S, Lee H, Wardlaw J. The Glymphatic System and Waste Clearance with Brain Aging: A Review. Gerontology. 2019;65(2):106-119. doi: 10.1159/000490349. Epub 2018 Jul 11. PMID 29996134
- [Background] Goodman JR, Adham ZO, Woltjer RL, Lund AW, Iliff JJ. Characterization of dural sinus-associated lymphatic vasculature in human Alzheimer's dementia subjects. Brain Behav Immun. 2018 Oct;73:34-40. doi: 10.1016/j.bbi.2018.07.020. Epub 2018 Jul 25. PMID 30055243
- [Background] MohanaSundaram A, Mofatteh M, Ashraf GM, Pratico D. Glymphotherapeutics for Alzheimer's disease: Time to move the needle. Ageing Res Rev. 2024 Nov;101:102478. doi: 10.1016/j.arr.2024.102478. Epub 2024 Aug 31. PMID 39222666
- [Background] Guo X, Zhang G, Peng Q, Huang L, Zhang Z, Zhang Z. Emerging Roles of Meningeal Lymphatic Vessels in Alzheimer's Disease. J Alzheimers Dis. 2023;94(s1):S355-S366. doi: 10.3233/JAD-221016. PMID 36683509
- [Background] Jiang H, Wei H, Zhou Y, Xiao X, Zhou C, Ji X. Overview of the meningeal lymphatic vessels in aging and central nervous system disorders. Cell Biosci. 2022 Dec 17;12(1):202. doi: 10.1186/s13578-022-00942-z. PMID 36528776
- [Background] Wu Y, Zhang T, Li X, Wei Y, Li X, Wang S, Liu J, Li D, Wang S, Ye T. Borneol-driven meningeal lymphatic drainage clears amyloid-beta peptide to attenuate Alzheimer-like phenotype in mice. Theranostics. 2023 Jan 1;13(1):106-124. doi: 10.7150/thno.76133. eCollection 2023. PMID 36593948
- [Background] Zhang X, Cao R, Zhu C, Yang L, Zheng N, Ji W, Liu P, Chi T, Ji X, Zheng Z, Chen G, Zou L. Mechanism of anti-AD action of OAB-14 by enhancing the function of glymphatic system. Neurochem Int. 2023 Oct 27:105633. doi: 10.1016/j.neuint.2023.105633. Online ahead of print. PMID 39491236
- [Background] Chen Y, He X, Cai J, Li Q. Functional aspects of the brain lymphatic drainage system in aging and neurodegenerative diseases. J Biomed Res. 2024 Mar 2;38(3):206-221. doi: 10.7555/JBR.37.20230264. PMID 38430054
- [Background] Pu T, Zou W, Feng W, Zhang Y, Wang L, Wang H, Xiao M. Persistent Malfunction of Glymphatic and Meningeal Lymphatic Drainage in a Mouse Model of Subarachnoid Hemorrhage. Exp Neurobiol. 2019 Feb;28(1):104-118. doi: 10.5607/en.2019.28.1.104. Epub 2019 Feb 28. PMID 30853828
- [Background] Li G, Cao Y, Tang X, Huang J, Cai L, Zhou L. The meningeal lymphatic vessels and the glymphatic system: Potential therapeutic targets in neurological disorders. J Cereb Blood Flow Metab. 2022 Aug;42(8):1364-1382. doi: 10.1177/0271678X221098145. Epub 2022 Apr 28. PMID 35484910
- [Background] Da Mesquita S, Louveau A, Vaccari A, Smirnov I, Cornelison RC, Kingsmore KM, Contarino C, Onengut-Gumuscu S, Farber E, Raper D, Viar KE, Powell RD, Baker W, Dabhi N, Bai R, Cao R, Hu S, Rich SS, Munson JM, Lopes MB, Overall CC, Acton ST, Kipnis J. Functional aspects of meningeal lymphatics in ageing and Alzheimer's disease. Nature. 2018 Aug;560(7717):185-191. doi: 10.1038/s41586-018-0368-8. Epub 2018 Jul 25. PMID 30046111
- [Background] Aspelund A, Antila S, Proulx ST, Karlsen TV, Karaman S, Detmar M, Wiig H, Alitalo K. A dural lymphatic vascular system that drains brain interstitial fluid and macromolecules. J Exp Med. 2015 Jun 29;212(7):991-9. doi: 10.1084/jem.20142290. Epub 2015 Jun 15. PMID 26077718